CLINICAL TRIAL: NCT05788536
Title: A PHASE 1/2, OPEN-LABEL, MULTICENTER TRIAL WITH A SINGLE ASCENDING DOSE COHORT WITH UNILATERAL INTRACOCHLEAR INJECTION FOLLOWED BY A BILATERAL INJECTION EXPANSION COHORT TO EVALUATE THE SAFETY, TOLERABILITY, AND EFFICACY OF DB-OTO IN CHILDREN AND INFANTS WITH BIALLELIC hOTOF MUTATIONS
Brief Title: A Study of DB-OTO, an Adeno-Associated Virus (AAV) Based Gene Therapy, in Children/Infants With Hearing Loss Due to Otoferlin Mutations
Acronym: CHORD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DB-OTO-001; 2022-000079-38 (EudraCT Number); 2024-511342-40-00 (EU CTIS Number)
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Congenital Hearing Loss Secondary to Biallelic Mutations of the Otoferlin Gene (OTOF)
Keywords: DB-OTO; Gene Therapy; Congenital Hearing Loss; Sensorineural Hearing Loss; Auditory Neuropathy; Pediatric; Cochlear Implant; Otoferlin; Deaf; Hard of hearing; Hearing impaired; Hearing disorder; Fully implantable hearing aid; Child; Infant; CHORD
MeSH Terms: conditions — Hearing Loss, Sensorineural; Auditory neuropathy; Deafness, Autosomal Recessive 9; Hearing Loss; Hearing Disorders

STUDY DESIGN:
Intervention Model Description: DB-OTO will be administered as a single intracochlear injection into one (Part A) or both ears (Part B). For bilateral injections (Part B), patients will receive DB-OTO in 1 surgical session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DB-OTO - Unilateral Dose Escalation (Experimental): Part A: Unilateral intracochlear dosing
  Interventions: Genetic: DB-OTO
- DB-OTO - Bilateral Dose Expansion (Experimental): Part B: Bilateral intracochlear dosing using the dose selected based on safety and efficacy data from Part A.
  Interventions: Genetic: DB-OTO

INTERVENTIONS:
Genetic: DB-OTO — DB-OTO will be administered as a single intracochlear injection into one ear (Part A).
  * LD Cohort (lower dose)
  * HD Cohort (high dose) - not implemented
  Arms: DB-OTO - Unilateral Dose Escalation
Genetic: DB-OTO — DB-OTO will be administered as a single intracochlear injection into both ears (Part B). For bilateral injections (Part B), patients will receive DB-OTO in 1 surgical session.
  Arms: DB-OTO - Bilateral Dose Expansion

SUMMARY:
Regeneron is conducting a study of an investigational new drug called DB-OTO. DB-OTO is a gene therapy that is being developed to treat children who have hearing loss due to changes in the otoferlin gene.

The purpose of this study is to:

* Learn about the safety of DB-OTO
* Determine how well DB-OTO is tolerated (does not cause ongoing discomfort)
* Evaluate the efficacy of DB-OTO (how well DB-OTO works)

DETAILED DESCRIPTION:
Former Sponsor Decibel Therapeutics

ELIGIBILITY:
Key Inclusion Criteria:

1. Willingness of at least 1 parent/legal guardian to provide written informed consent (and patient to provide assent, when applicable) and willingness to comply with trial protocol; to consent to genetic testing for the patient (and patient to provide assent, when applicable) in order to evaluate a panel of hearing loss-related genes; and to consent to vaccinations for the patient (and patient to provide assent, when applicable) in accordance with the country-specific pediatric immunization schedule as described in the protocol
2. Patient is aged <18 years and able to perform all necessary assessments to qualify for enrollment and dosing in the corresponding cohort at the time the parent/legal guardian signing the informed consent form (and patient providing assent, when applicable)
3. Presence of biallelic, likely pathogenic or pathogenic OTOF variants
4. No clinically significant laboratory findings on clinical laboratory tests at time of Screening as described in the protocol
5. Audiological Criteria:

   1. Investigator diagnoses the patient with profound sensorineural hearing loss (SNHL; ≥90 dB HL) based on behavioral and physiologic measurements (ABR) of inner ear function
   2. Outer hair cell presence is confirmed via presence of otoacoustic emissions (≥6 dBSNR) at ≥3 frequencies from 1 to 8 kHz in the ear(s) to be injected with DB-OTO. Alternatively, for children >24 months to <18 years of age, outer hair cell presence can be confirmed via presence of the cochlear microphonic in the ear(s) to be injected with DB-OTO.
6. No evidence from measures of hearing loss that show a dependence on body temperature
7. From study start and for the duration of the short-term follow-up period (48 weeks): Female patients of childbearing potential and fertile males, must agree to use highly effective contraception. Female patients must agree not to become pregnant. Fertile male patients must agree not to father a child or donate sperm, for 48 weeks and in cases of early withdrawal, for at least 12 months after DB-OTO administration.

Key Exclusion Criteria:

1. History of prior treatment with gene therapy
2. Surgical anatomy that would preclude or meaningfully impact the planned surgical approach as indicated by medical imaging (eg, computed tomography [CT] or magnetic resonance imaging [MRI]) in the ear(s) to be injected with DB-OTO
3. History or presence of other permanent or untreatable hearing loss conditions
4. Prior or current history of malignancies
5. Prior or current history of meningitis
6. History or presence of cochlear implants in the ear(s) to be injected with DB-OTO
7. History of risk factor(s) for auditory neuropathy not caused by OTOF pathogenic variants including but not limited to: prematurity, low birth weight, hyperbilirubinemia, neonatal intensive care unit (NICU) admission, and/or low Apgar scores as described in the protocol

Note: Other protocol-defined inclusion/exclusion criteria apply

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2031-04-19 (Estimated); Study Completion 2031-04-19 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | Up to week 48
Achievement of a hearing sensitivity threshold of ≤70 dB assessed by average pure tone audiometry (PTA) | Up to week 48

SECONDARY OUTCOMES:
Auditory Brainstem Response (ABR) to click | Up to week 48
Achievement of a hearing sensitivity threshold of ≤45 dB assessed by average PTA | Up to week 48
Achievement of hearing sensitivity threshold of ≤25 dB assessed by average PTA | Up to week 48
Speech perception scores by age-appropriate tests | Up to week 48
Speech Awareness Threshold (SAT): achievement of a threshold of ≤70 dB | Up to week 48
SAT: achievement of a threshold of ≤45 dB | Up to week 48
SAT: achievement of threshold of ≤25 dB | Up to week 48
Speech Reception Threshold (SRT): achievement of a threshold of ≤70 dB | Up to week 48
SRT: achievement of a threshold of ≤45 dB | Up to week 48
SRT: achievement of a threshold of ≤25 dB | Up to week 48
Severity in speech perception ability assessed by Global Impression scales, determined by clinician | Up to week 48
Severity in speech perception ability assessed by Global Impression scales, determined by parent/legal guardian | Up to week 48
Change in speech perception ability assessed by Global Impression scales, determined by clinician | Up to week 48
Change in speech perception ability assessed by Global Impression scales, determined by parent/legal guardian | Up to week 48
Average PTA threshold in the subset of patients who achieved an average PTA threshold ≤70 dB | Up to week 48
Average PTA threshold in the subset of patients who achieved an average PTA threshold >70 dB but ≤85 dB | Up to week 48
Achievement of a hearing sensitivity threshold improvement of ≥10 dB from baseline | Up to week 48
Time to an average PTA threshold ≤70 dB | Up to week 48
Incidence of patients who regress to >70 dB after having achieved average PTA threshold ≤70 dB | Up to week 48
Persistence of an average PTA threshold ≤70 dB | Up to week 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (15):
- United States (9):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Nemours Children s Clinic, Jacksonville, Florida
  - Nemours Childrens Hospital, Orlando, Florida
  - Boston Children's Hospital - Main, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University Hospital Tubingen, Tübingen, Germany
- Spain (3):
  - Hospital Universitario Materno Infantil en las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Ramon y Cajal University Hospital, Madrid
  - Clinica Universidad de Navarra- Pamplona, Pamplona
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge University Hospitals NHS FT, Cambridge
  - Great Ormond Street Hospital For Children NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Valayannopoulos V, Bance M, Carvalho DS, Greinwald JH Jr, Harvey SA, Ishiyama A, Landry EC, Lowenheim H, Lustig LR, Manrique M, Nash R, Polo R, Pritchett CV, Rubinstein JT, Shearer AE, Del Castillo I, Anderson JJ, Corrales CE, Quigley TM, Riggs WJ, Weber P, Wilson G, Irvin SC, Hassan HE, Chen Y, Liu R, Drummond MC, Sabin LR, Musser BJ, Yancopoulos GD, Kyratsous CA, Herman GA, Baras A, Whitton JP; CHORD Study Group. DB-OTO Gene Therapy for Inherited Deafness. N Engl J Med. 2025 Oct 12. doi: 10.1056/NEJMoa2400521. Online ahead of print. PMID 41085057
- See also: Patients, Caregivers & HCPs: Contribute to Genetic Hearing Loss Research — https://portal.sanogenetics.com/study/genetic-hearing-loss-trials